CLINICAL TRIAL: NCT06792435
Title: A Phase I/Ⅱ, First-in-Human Study of XNW27011 in Patients with Locally Advanced And/or Metastatic Solid Tumors
Brief Title: XNW27011 Study of Advanced Solid Tumor Subjects Who Failed Standard Therapies.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XNW27011-I/II-01
Record Dates: First submitted 2024-12-25; First posted 2025-01-24 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Adenocarcinoma Metastatic; Lung Cancer (NSCLC); Ovarian Cancer; Colorectal Cancer Metastatic; Biliary Tract Cancer; Gastric Carcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Biliary Tract Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I Dose Escalation (Experimental): Based on the preclinical data of XNW27011, the dose-escalation study will start from the initial dose of 0.6 mg/kg. Dose escalation will be performed by using a modified Fibonacci method with a slightly fine-tuned dose escalation amplitude. The first two dose escalations will be by 100% of the preceding dose and thereafter by 50%, 33%, 25% and 25% of the preceding doses. Therefore, there are 7 dose cohorts for projected dose escalations as follows
  Interventions: Drug: XNW27011
- Phase II: Expanded cohorts (Experimental): The SRC will select up to 3 recommended doses for Phase II study based on the safety, PK, ADA and preliminary efficacy data from Phase I study (dose escalation). Phase Ⅱwill include 4 patient groups, and up to 3 dose cohorts for each patient group. Approximately 20 Chinese or U.S. patients will be enrolled to each dose cohort with an approximately total of 240 patients in the Phase II study to further evaluate the antitumor activity, safety, tolerability, PK and incidence of ADA for XNW27011.
  Interventions: Drug: XNW27011

INTERVENTIONS:
Drug: XNW27011 — Eligible patient(s) in each dose cohort will receive the assigned XNW27011 dose administration every 3 weeks (Q3W, cycle) until intolerable toxicity, progression of the disease without clinical benefit, or withdrawal of informed consent.
  An accelerated titration scheme will be used for the first two dose levels (0.6 mg/kg and 1.2 mg/kg) starting from 0.6 mg/kg dose as follows:
  The first patient will be enrolled for 0.6 mg/kg dose. If the subject shows no significant toxicity in cycle 1 (DLT observation period), the second patient will be enrolled for 1.2 mg/kg.
  3 + 3 dose escalation:3 patients will be enrolled to the dose cohort first，If 1 of 3 patients experiences a DLT, up to 3 more patients will be enrolled in the same dose cohort.. If none of the additional 3 patients experiences a DLT, dose escalation will continue to the next dose.Dose escalation will be stopped when 2 or more patients out of 3 to 6 patients at the same dose level experience a DLT.
  Arms: Phase I Dose Escalation
Drug: XNW27011 — Group A: Gastric/gastroesophageal junction adenocarcinoma with CLDN18.2 expression, tentatively expand with 3.6, 3.0, 2.4 mg/kg. Group B: Pancreatic adenocarcinoma with CLDN18.2 expression, tentatively expand with 3.6, 3.0, 2.4 mg/kg. Group C: Ovarian cancer with CLDN18.2 expression, tentatively expand with 3.6, 3.0, 2.4 mg/kg. Group D: Other tumors with CLDN18.2 expression, including but not limited to esophagus adenocarcinoma, lung cancer, colorectal cancer, and biliary tract cancer,tentatively expand with 3.6, 3.0, 2.4 mg/kg.
  Arms: Phase II: Expanded cohorts

SUMMARY:
This is a global, multi-center, open-label, Phase I/II first-in-human study of XNW27011 monotherapy as an investigational product (IP) in patients with locally advanced and/or metastatic solid tumors who have failed or are intolerant to standard therapies. XNW27011 is an antibody-drug conjugate (ADC) targeting Claudin 18.2 (CLDN18.2), a transmembrane protein important to tight junctions. The study consists of 2 parts: Part 1 is the dose-escalation phase (Phase I), and Part 2 is the does-expansion phase (Phase II). In phase I part of the study, approximately 42 patients with locally advanced and/or metastatic solid tumors will be enrolled, irrespective of CLDN18.2 expression. However, the most recently available tumor tissue specimen will be collected (if available) for a retrospective CLDN18.2 expression confirmation. In phase II part of the study, only patients with confirmed CLDN18.2 expression by IHC in the central laboratory will be enrolled.The phase II part of the study will consist of the following four groups，Up to three dose cohorts for each patient group are planned currently. Each dose cohort will include approximately 20 patients. Approximately 240 patients evaluable will be enrolled in Phase Ⅱ part of the study.

DETAILED DESCRIPTION:
This is a global, multi-center, open-label, Phase I/II first-in-human study of XNW27011 monotherapy as an investigational product (IP) in patients with locally advanced and/or metastatic solid tumors who have failed or are intolerant to standard therapies. XNW27011 is an antibody-drug conjugate (ADC) targeting Claudin 18.2 (CLDN18.2), a transmembrane protein important to tight junctions. The study consists of 2 parts: Part 1 is the dose-escalation phase (Phase I), and Part 2 is the does-expansion phase (Phase II). In phase I part of the study, approximately 42 patients with locally advanced and/or metastatic solid tumors will be enrolled, irrespective of CLDN18.2 expression. However, the most recently available tumor tissue specimen will be collected (if available) for a retrospective CLDN18.2 expression confirmation. In phase II part of the study, only patients with confirmed CLDN18.2 expression by IHC in the central laboratory will be enrolled.The phase II part of the study will consist of the following four groups，Up to three dose cohorts for each patient group are planned currently. Each dose cohort will include approximately 20 patients. Approximately 240 patients evaluable will be enrolled in Phase Ⅱ part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Phase I (Dose Escalation)：

  1. Patients are willing and able to provide written informed consent or where consent is provided by legally authorized representatives.
  2. Age ≥18 years old when signing the informed consent form.
  3. Patients with a histologically or cytologically-confirmed, locally advanced or metastatic solid tumor, which has failed on standard therapy or is intolerable to available standard therapy, or there is no available standard therapy for the tumor. The advanced solid tumors include but are not limited to gastric and gastroesophageal junction adenocarcinoma, pancreatic adenocarcinoma, esophageal adenocarcinoma, ovarian cancer, lung cancer, colorectal cancer, andbiliary tract cancer.
  4. The enrollment is not restricted to patients with tumor expressing CLDN18.2. However patients are required to provide tumor tissue sections for CLDN18.2 expression confirmation.
  5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
  6. Estimated life expectancy > 12 weeks.
  7. At least one measurable cancer lesion as defined by the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
  8. Adequate organ function, evidenced by the following laboratory results:

     1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
     2. Platelet count ≥ 100 × 109/L.
     3. Hemoglobin ≥ 9.0 g/dL.
     4. Total bilirubin ≤ 1.5 × the upper limit of normal (ULN).
     5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 × ULN (if liver metastases are present, ≤ 3 × ULN).
     6. Creatinine clearance (Ccr) ≥60 mL/minute as calculated using themodified Cockcroft-Gault equation.
     7. QTc prolongation to ≤480 milliseconds (ms) (based on the average of 3 screening electrocardiograms) (QTc interval corrected by Fridericia's Correction Formula, QTcF = QT/(RR0.33).
     8. Echocardiographic LVEF (left ventricular ejection fraction) ≥ 50%.
  9. Female patients of childbearing potential, who are willing to use a highly effective method of birth control during the study, and for at least 180 days after the last dose of study medication.

     1. Childbearing potential is defined as any female who has experienced menarche and does not meet the criteria for postmenopausal, which is defined as the past 12 months with no menses without an alternative medical cause or permanently sterilized (e.g., has undergone bilateral tubal occlusion/ligation, hysterectomy, bilateral oophorectomy, bilateral salpingectomy).
     2. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, or a vasectomized partner.
  10. Male patients with female sexual partners of childbearing potential are eligible for inclusion if they agree to use medically acceptable birth control during the study, and for 180 days after the last dose of study medication. Sexual abstinence, vasectomy, or a condom used with a spermicide are medically acceptable birth control methods for males. Male subjects must agree not to donate sperm for a period of 180 days after the last dose of study treatment.

PHASE Ⅱ (DOSE EXTENSION)：

1. Subjects are willing and able to provide written informed consent or where consent is provided by legally authorized representatives.
2. Age ≥18 years old when signing the informed consent form.
3. Patients with histologically or cytologically confirmed, locally advanced or metastatic solid tumors, which have failed on standard therapy, or are intolerable to available standard therapy, or for which there is no available standard therapy.

   Patients are grouped by anatomic locations of solid tumors:

   Group A: gastric adenocarcinoma/gastroesophageal junction adenocarcinoma. Group B: pancreatic adenocarcinoma. Group C: ovarian cancer. Group D: other cancer including esophagus adenocarcinomas, lung cancer, colorectal cancer, and biliary tract cancer.
4. Only patients with tumor expressing CLDN 18.2 will be enrolled. The most recently available tumor samples of patients will be examined by IHC at a central laboratory. If no archived tumor samples are available or the archived tumor samples are deemed to be inappropriate for the confirmation of CLDN18.2 expression, a new biopsy must be performed to obtain the tumor sample to confirmation of CLDN18.2 expression.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Estimated life expectancy > 12 weeks.
7. At least one measurable cancer lesion as defined by the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1).
8. Adequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
   2. Platelet count ≥ 100 × 109/L.
   3. Hemoglobin ≥ 9.0 g/dL.
   4. Total bilirubin ≤ 1.5 × the upper limit of normal (ULN).
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5× ULN (if liver metastases are present, ≤ 3 × ULN).
   6. Creatinine clearance (Ccr) ≥50 mL/minute as calculated using the modified Cockcroft-Gault equation.
   7. QTc prolongation to ≤ 480 millisecond (ms) (based on the average of 3 screening electrocardiograms) (QTc interval corrected by Fridericia's Correction Formula, QTcF = QT/(RR0.33).
   8. Echocardiographic LVEF (left ventricular ejection fraction) ≥ 50%.
9. Female patients of childbearing potential, who are willing to use a highly effective method of birth control during the study and for at least 180 days following the last dose of study medication.

   1. Childbearing potential is defined as any female who has experienced menarche and does not meet the criteria for postmenopausal, which is defined as the past 12 months with no menses without an alternative medical cause or permanently sterilized (e.g., has undergone bilateral tubal occlusion/ligation, hysterectomy, bilateral oophorectomy, bilateral salpingectomy).
   2. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence, or a vasectomized partner.
10. Male patients with female sexual partners of childbearing potential are eligible for inclusion if they agree to use medically acceptable birth control for 180 days following the last dose of study medication. Sexual abstinence, vasectomy, or a condom used with a spermicide are medically acceptable birth control methods for males. Male subjects must agree not to donate sperm for a period of 180 days after the last dose of study treatment.

Exclusion Criteria:

* PHASE I (DOSE ESCALATION)：

  1. Prior severe allergic reaction or intolerance to a monoclonal antibody, including humanized or chimeric antibodies.
  2. Prior severe allergic reaction or intolerance to the Topoisomerase I Inhibitor or Topoisomerase Inhibitor-Based ADC (e.g: Fam-trastuzumab deruxtecan-nxki, Sacituzumab govitecan-hziy, Irinotecan, Topotecan) or any excipient in the XNW27011 formulation.
  3. Having any of the following medical conditions in the past or at present:

     1. Acquired or congenital immunodeficiency diseases or organ transplantation.
     2. Past myocardial infarction (within 6 months before the first administration), hospitalization for congestive heart failure within 12 months before the first administration, severe or unstable angina, coronary or peripheral artery bypass grafting, New York Heart Association (NYHA) grade Ⅲ or IV heart failure, uncontrollable hypertension (Systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg at rest).
     3. Concomitant diseases that will seriously endanger the safety of the subject or affect the completion of the tests, such as active gastrointestinal bleeding, active peptic ulcer, intestinal obstruction, intestinal paralysis, interstitial pneumonia, lung fibrosis, kidney failure, and uncontrolled diabetes(HbA1c>8%).
     4. History of or currently suffering from uncontrolled primary or metastasized brain tumors, except that the investigator believes that the disease has been stabilized in patients, or whose local treatment has ended.
     5. History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of the XNW27011.
     6. Past or current mental illness that is difficult to control.
     7. Human immunodeficiency virus (HIV) infection, syphilis infection, or active hepatitis B or C infection. Note: Syphilis infection refers to active syphilis or latent syphilis that requires treatment.
     8. Patients who have active infections that required systemic treatment within 2 weeks prior to the first dose of XNW27011.
     9. Clinically significant third spacing (large amount of pleural fluid or ascites, judged by treating physician) that is uncontrollable by drainage or other methods.
     10. Having any adverse event from prior anti-tumor treatments that have not yet recovered to Grade 0 or 1 per NCI-CTCAE v5.0 (except alopecia).
  4. History of treatment:

     1. Patients who have previously participated in clinical trials of other drugs within 4 weeks before the first dose of XNW27011.
     2. Received anti-tumor therapy (chemotherapy, radiotherapy, immunologic therapy or biological therapy,) within 3 weeks, prior to the first dose of XNW27011, or received small molecular targeted therapy, anti-tumor medicinal herb or proprietary Chinese traditional medicines within 2 weeks, or received palliative radiotherapy for bone metastases within 2 weeks, or received nitrosoureas or mitomycin C within 6 weeks.
     3. Received major surgical or interventional treatment within 4 weeks prior to the first dose of XNW27011, with the exception of tumor biopsy, puncture, etc.
     4. Received systemic steroid therapy for a long period of time (≥20 mg of prednisone/day or equivalent for >7 days). (Short-term use of no more than 7 days or steroid therapy withdrawal longer than 2 weeks prior to the first dose of XNW27011 can be selected).
     5. Received live vaccines within 4 weeks prior to the first dose of XNW27011 or plan to take any live vaccine during the study period.
     6. Received strong inhibitors or inducers of CYP3A4, or strong inhibitors of CYP2D6 within 2 weeks or five half-lives (whichever is shorter) of the inhibitor or inducer prior to the first dose of XNW27011.
  5. Women who are pregnant or breastfeeding, or women whose serum pregnancy test results are positive during the screening period (female patients who are infertile do not need to undergo a pregnancy test, e.g., female patients who underwent hysterectomy, bilateral tubal occlusion/ ligation, bilateral salpingectomy, or bilateral oophorectomy in the past, or women with resection or amenorrhea ≥12 months).
  6. Patients who have poor compliance and are not expected to cooperate to complete the study procedures, or who are deemed unsuitable to participate in the clinical research by the investigator. PHASE Ⅱ (DOSE EXTENSION)：

  <!-- -->

  1. Prior severe allergic reaction or intolerance to a monoclonal antibody, including humanized or chimeric antibodies.
  2. Prior severe allergic reaction or intolerance to the Topoisomerase I Inhibitor or Topoisomerase Inhibitor-Based ADC (e.g: Fam-trastuzumab deruxtecan-nxki, Sacituzumab govitecan-hziy, Irinotecan, Topotecan) or any excipient in the XNW27011 formulation.
  3. Having any of the following medical conditions in the past or present:

     1. Acquired or congenital immunodeficiency diseases or organ transplantation.
     2. Past myocardial infarction (within 6 months before the first administration), hospitalization for congestive heart failure within 12 months before the first administration, severe or unstable angina, coronary or peripheral artery bypass grafting, New York Heart Association (NYHA) grade Ⅲ or IV heart failure, uncontrollable hypertension (Systolic BP ≥ 160 mmHg and/or diastolic BP ≥ 100 mmHg at rest).
     3. Concomitant diseases that will seriously endanger the safety of the subject or affect the completion of the study, such as active gastrointestinal bleeding, active peptic ulcer, intestinal obstruction, intestinal paralysis, interstitial pneumonia, lung fibrosis, kidney failure, and uncontrolled diabetes (HbA1c>8%).
     4. Previously or currently suffering from uncontrollable primary or metastasized brain tumors, except that the investigator believes that the disease has been stabilized in patients, or whose local treatment has ended.
     5. History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of XNW27011.
     6. Past or current mental illness that is difficult to control.
     7. Human immunodeficiency virus (HIV) infection, syphilis infection, or active hepatitis B or C infection.

        Note: Syphilis infection refers to active syphilis or latent syphilis that requires treatment.
     8. Patients who have active infections that required systemic treatment within 2 weeks prior to the first dose of XNW27011.
     9. Has multiple primary malignancies within 5 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, and other solid tumors curatively treated.
     10. Clinically significant third spacing (large amount of pleural fluid or ascites, judged by treating physician) that is uncontrollable by drainage or other methods.
     11. Having any adverse event from prior anti-tumor treatments that have not yet recovered to Grade 0 or 1 per NCI-CTCAE v5.0 (except alopecia).
  4. History of treatment:

     1. Patients who have previously been treated with ADCs or CAR-T targeting CLDN18.2, or participated in clinical trials of other drugs within 4 weeks before the first dose of XNW27011.
     2. Received anti-tumor therapy (chemotherapy, radiotherapy, immunologic therapyor biological therapy) within 3 weeks, prior to the first dose of XNW27011, or received small molecular targeted therapy, anti-tumor medicinal herb or proprietary Chinese traditional medicines within 2 weeks, or received palliative radiotherapy for bone metastases within 2 weeks, or received nitrosoureas or mitomycin C within 6 weeks.
     3. Have received major surgical or interventional treatment within 4 weeks prior to the first dose of XNW27011, with the exception for tumor biopsy, puncture, etc.
     4. Received systemic steroid therapy for a long period of time (≥20 mg of prednisone/day or equivalent for >7 days). (Short-term use of no more than 7 days or steroid therapy withdrawal longer than 2 weeks prior to the first dose of XNW27011 can be selected).
     5. Received live vaccines within 4 weeks prior to the first dose of XNW27011or planned to take any live vaccine during the study period.
     6. Received strong inhibitors or inducers of CYP3A4, or strong inhibitors of CYP2D6 within 2 weeks or five half-lives (whichever is shorter) of the inhibitor or inducer prior to the first dose of XNW27011.
  5. Women who are pregnant or breastfeeding, or women whose serum pregnancy test results are positive during the screening period (female patients who are infertile do not need to undergo a pregnancy test, e.g., female patients who underwent hysterectomy, bilateral tubal occlusion/ligation, bilateral salpingectomy, or bilateral oophorectomy in the past and women with resection or amenorrhea ≥12 months).
  6. Patients who have poor compliance and are not expected to cooperate to complete the study procedures, or who are deemed unsuitable to participate in the clinical research by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I (Dose Escalation):To determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of XNW27011 | Baseline up to approximately 2 years
  In the dose escalation phase, if there are ≥ 2 cases of DLT among 3-6 subjects at a dose level during the DLT observation period (Cycle 1, 21days), the previous dose or intermediate dose (the midway dose between the previous dose group and the intolerant dose group) may be defined as MTD.
Phase Ⅱ (Dose Expansion):To evaluate the objective response rate (ORR) of XNW27011 by cohorts at RP2D. The objective response includes the complete response (CR) and the partial response (PR). | Baseline up to approximately 2 years
  To evaluate the objective response rate (ORR) of XNW27011 by cohorts at RP2D. The objective response includes the complete response (CR) and the partial response (PR).

SECONDARY OUTCOMES:
Phase I (Dose Escalation):To assess the dose limiting toxicities (DLTs) of XNW27011 when administered intravenously (IV) as a monotherapy during the first cycle (3 weeks [21 days]) to patients with locally advanced and/or metastatic solid tumors. | 3 weeks
  To assess the dose limiting toxicities (DLTs) of XNW27011 when administered intravenously (IV) as a monotherapy during the first cycle (3 weeks [21 days]) to patients with locally advanced and/or metastatic solid tumors.
Phase I (Dose Escalation)：To assess the overall safety of XNW27011 when administered IV as a monotherapy every cycle (3 weeks [Q3W]) to patients with locally advanced and/or metastatic solid tumors. | 3 weeks
  The incidence and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Phase I (Dose Escalation)：To assess the pharmacokinetic (PK) profiles of XNW27011, total antibody (XNW27011-TAb, including conjugated and unconjugated), the topoisomerase I inhibitor YL0010014 (payload/toxin) and the major metabolites. | Baseline up to approximately 2 years
  To assess the pharmacokinetic (PK) profiles of XNW27011, total antibody (XNW27011-TAb, including conjugated and unconjugated), the topoisomerase I inhibitor YL0010014 (payload/toxin) and the major metabolites.
Phase I (Dose Escalation)：To evaluate the preliminary efficacy of XNW27011 as a monotherapy. | Baseline up to approximately 2 years
  According to RECIST 1.1, the proportion of subjects' ORR was evaluated by researchers.
Phase I (Dose Escalation)：To assess the incidence of anti-drug antibody (ADA) against XNW27011. | Baseline up to approximately 2 years
  To assess the incidence of anti-drug antibody (ADA) against XNW27011.
Phase I (Dose Escalation)：To assess the relationship between claudin 18.2 (CLDN18.2) expression and the antitumor response of XNW27011. | Baseline up to approximately 2 years
  According to the expression rate of claudin 18.2 and the corresponding best ORR, the influence of claudin 18.2 expression rate on the curative effect was analyzed.
Phase Ⅱ (Dose Expansion)：To assess the safety of XNW27011 at the RP2D. | Baseline up to approximately 2 years
  The incidence and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Phase Ⅱ (Dose Expansion)：To evaluate the efficacy of XNW27011 at the RP2D： Disease control rate (DCR) | Baseline up to approximately 2 years
  DCR is defined as the percentage of subjects with the best tumor evaluation of CR, PR or SD among all patients with measurable disease at baseline.
Phase Ⅱ (Dose Expansion)：To evaluate the efficacy of XNW27011 at the RP2D：Duration of response (DOR) | Baseline up to approximately 2 years
  DOR is defined as the duration from the first documentation of disease response (CR/PR) to the first documentation of disease progression or death; the end date is the same as the date of disease progression defined for PFS or death due to any cause, the start date is the date of the first evaluation of PR or CR.
Phase Ⅱ (Dose Expansion)：To evaluate the efficacy of XNW27011 at the RP2D：Time to response (TTR) | Baseline up to approximately 2 years
  TTR is defined as the time from the date of first dose to the date of first meeting response criteria.
Phase Ⅱ (Dose Expansion)：To evaluate the efficacy of XNW27011 at the RP2D：Progression-Free Survival (PFS) | Baseline up to approximately 2 years
  PFS is defined as the length of time from the first dose to progression of disease or death.
Phase Ⅱ (Dose Expansion)：To evaluate the efficacy of XNW27011 at the RP2D：Overall survival (OS) | Baseline up to approximately 2 years
  OS is defined as the time from the date of first dose to the date of death due to any cause.
To assess the relationship between CLDN18.2 expression and the antitumor response of XNW27011. | Baseline up to approximately 2 years
  According to the expression rate of claudin 18.2 and the corresponding best ORR, the influence of claudin 18.2 expression rate on the curative effect was analyzed.
To assess the incidence of ADA against XNW27011. | Baseline up to approximately 2 years
  To assess the incidence of ADA against XNW27011.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No